CLINICAL TRIAL: NCT04699942
Title: Pilot Study to Evaluate the Revoxa™ System in Hypoxic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. David Maslove (Other)
Collaborators: Ironstone Professional Development (Unknown)
Responsible Party: Sponsor-Investigator, Dr. David Maslove, Associate Professor, Queen's University
Organization: Queen's University (Other)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 6031410
Record Dates: First submitted 2021-01-05; First posted 2021-01-07 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Hypoxemia
Keywords: hypoxia; hypoxemia; oxygen delivery; COVID-19; rebreather circuit
MeSH Terms: conditions — Hypoxia; COVID-19

STUDY DESIGN:
Intervention Model Description: Following baseline measurement, either conventional low-flow oxygen delivery or oxygen delivery via the Revoxa Oxygen Rebreather device is initiated for 20 minutes, followed by the other modality for 20 minutes. The order of treatments will be determined quasi-randomly based on whether the patient is enrolled on an odd-numbered day, or an even-numbered day.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional (Active Comparator): Conventional low-flow Oxygen Delivery
  Interventions: Device: Conventional (low flow) oxygen delivery via nasal cannula
- Revoxa (Experimental): Oxygen Delivery via Revoxa Oxygen Rebreather Device
  Interventions: Device: Revoxa Oxygen Rebrearther

INTERVENTIONS:
Device: Conventional (low flow) oxygen delivery via nasal cannula — Conventional (low flow) oxygen delivery via nasal cannula or face mask for 20 minutes
  Arms: Conventional
Device: Revoxa Oxygen Rebrearther — Oxygen delivery via Revoxa Oxygen Rebreather device for 20 minutes
  Arms: Revoxa

SUMMARY:
Patients with COVID-19 may suffer from profound hypoxia, requiring the use of supplemental oxygen at high concentrations and flow rates. Non-invasive oxygen delivery systems such as high-flow nasal cannula and non-invasive ventilation have been used in an attempt to avoid the need for intubation and invasive mechanical ventilation. These systems consume large amounts of oxygen, which prevents them from being used in areas without high pressure oxygen sources. In addition, they generate aerosols which have the potential to spread infectious pathogens from the patient's respiratory tract to healthcare workers or other patients in the environment. This study aims to investigate a computer controlled rebreather system which functions to maintain a high fraction of inspired oxygen while minimizing the production of aerosol, among hospitalized patients requiring respiratory support due to hypoxemia. The Revoxa Oxygen Rebreather device can reduce the amount of wasted oxygen and can reduce the potential for any exhaled pathogens entering the surroundings. This type of breathing device is a promising oxygen delivery treatment, but it is not clear if it can offer comparable results to standard treatment. The purpose of this study is to compare the Revoxa Oxygen Rebreather device to standard oxygen delivery methods, including nasal cannula and face mask oxygen, in order to see if similar oxygenation can be achieved at comparable or lower rates of oxygen usage.

DETAILED DESCRIPTION:
This study aims to investigate a two-phase rebreather system (Revoxa Oxygen Rebreather device) among hospitalized patients requiring oxygen therapy. This system can deliver a high fraction of inspired oxygen (FiO2) using a very low flow oxygen source with reduced or no aerosolization. This could provide effective respiratory support with reduced waste and risk of spreading of infectious particles. Such a device could also be used in field hospitals and other makeshift care centers in the event of a surge in demand, because it obviates the need for the type of high-flow oxygen infrastructure that is typically limited to hospital settings.

This is a prospective comparative study of sequential interventions to evaluate the ability of the Revoxa Oxygen Rebreather device (RO) to improve and maintain oxygen saturation at satisfactory levels compared to conventional low-flow supplemental oxygen delivery (COD) via nasal cannula or face mask. Prior to conducting study procedures in the patient population, feasibility of trial procedures will be determined among 3 healthy adults (Group A). The initial procedural test in a healthy sample will not be included in the endpoint assessment. Following initial trial conduct in a healthy sample, 20 adult patients requiring supplemental oxygen will be recruited: adults with non-severe hypoxemia (Group B), followed by enrollment of adults with hypoxemia of any severity not requiring mechanical ventilation (Group C). Baseline measures of oxygen saturation, oxygen flow rate, vital signs (respiratory rate, heart rate, and blood pressure), and patient self-reported dyspnea and comfort will be recorded prior to initiating treatment. Following baseline measurement, either conventional low-flow oxygen delivery or oxygen via the Revoxa Oxygen Rebreather device will be initiated for 20 minutes, followed by the other modality for 20 minutes. To avoid any bias that may be introduced by a fixed sequence of device utilization (eg. COD, then RO), the order in which devices are used will be determined quasi-randomly based on whether the patient is enrolled on an odd numbered day, or an even numbered day. Vital signs, supplemental oxygen, and self-reported dyspnea measures are captured during both treatment regimens. Participants may verbally withdraw at any time by contacting one of the clinical or research staff. At that point, all data collection relating to the withdrawn study participant will be terminated. If the participant wishes, all existing data will be deleted (with the exception of the signed consent form and data related to the consent withdrawal - including the reason for the withdrawal). Additional participants will be recruited to maintain an adequate sample size in the event that participants are withdrawn from the study.

ELIGIBILITY:
Inclusion Criteria:

Group A - Healthy adults (≥ 18 years of age) with SpO2 ≥ 96% without oxygen supplementation

Group B - non-severe hypoxemia requiring supplemental oxygen as defined by:

* SpO2 > 96% with oxygen face mask or nasal cannula with low flow oxygen <5LPM
* Adults (≥ 18 years of age)

Group C - Hypoxemia requiring supplemental oxygen as defined by:

* Oxygen saturation (SpO2) ≤ 92% on room air as measured by pulse oximetry; or
* SpO2 < 94% with oxygen face mask or nasal cannula with low flow oxygen <5LPM
* Adults (≥ 18 years of age)

Exclusion Criteria:

* Acute / unstable cardiovascular condition
* Pregnancy
* Imminent need for intubation or noninvasive ventilation
* Glasgow coma scale <14

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Oxygen flow required to achieve SpO2 >96%. | Baseline to 20 minutes
  Oxygen flow required to achieve SpO2 >96%.

SECONDARY OUTCOMES:
Average oxygen consumption | Baseline to 20 minutes
  Average oxygen consumption
Peak SpO2 | Baseline to 20 minutes
  Peak SpO2
Patient-reported dyspnea (Modified Borg Scale) | Baseline to 20 minutes
  Patient-reported dyspnea (Modified Borg Scale)
Patient-reported comfort (Visual Analogue Scale) | Baseline to 20 minutes
  Patient-reported comfort (Visual Analogue Scale)

CONTACTS AND LOCATIONS:
Locations (1):
- Kingston Health Sciences Centre, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No